CLINICAL TRIAL: NCT00376649
Title: Development of Workshop for Lifestyle Changing for Crohn's Disease Patients and Its Affect on the Disease's Indexes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding was not granted
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 16-031106-HMO-CTIL
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Crohn's Disease
Keywords: crohns; quality of life; lifestyle changing; remmision
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Behavioral: lifestyle changing workshop

SUMMARY:
Subjects that participate in the practical workshop will improve their quality of life and will stay longer in remmision , in compare to the participants that will continue their regular threatment

DETAILED DESCRIPTION:
Participants will be randomly assigned to a regular threatment (control group) or to a lifestyle changing workshop. The workshop will consist of 11 meetings with behavioral lessons in nutrition, cooking, stress realese and physical activity. The study population will include 100 crohn's disease patients in remmision that will be recruited and will be randomly divided into two groups: an intervention group of 50 will commence the workshop during 2007 and a control group of 50 who will continue their regular threatment. an IBDQ , CDAI and blood samples for metabolic index will be taken from the participant in the staudy before entering the study and every half a year for three years.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* diagnosed with CD
* Crohn's Disease Activity Index (CDAI) of under 170
* a minimum of 75% of the meetings

Exclusion Criteria:

* patients with a stoma
* and patients with a planned admission to the hospital for surgery or other treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rifat safadi, md, Principal Investigator — hadassah univercity hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel